CLINICAL TRIAL: NCT00622648
Title: International, Multi-center, Randomized, Double Blind Study to Compare the Overall Mortality in Acutely Ill Medical Patients Treated With Enoxaparin Versus Placebo in Addition to Graduated Elastic Stockings
Brief Title: Study to Evaluate the Mortality Reduction of Enoxaparin in Hospitalized Acutely Ill Medical Receiving Enoxaparin
Acronym: LIFENOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENOXA_C_01249
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Acute Illness
Keywords: Medical prevention therapy
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental): Enoxaparin: 40 mg once daily for 6 to 14 days (10 ± 4 days)
  Interventions: Drug: Enoxaparin
- B (Placebo Comparator): Enoxaparin placebo 40mg once daily for 6 to 14 days (10 ± 4 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enoxaparin — 40 mg once daily for 6 to 14 days (10 ± 4 days)
  Arms: A
Drug: Placebo — Enoxaparin placebo 40mg once daily for 6 to 14 days (10 ± 4 days)
  Arms: B

SUMMARY:
The primary objective:

* To demonstrate in patients hospitalized for an acute medical illness that enoxaparin with Graduated Elastic Stockings is superior to enoxaparin-placebo with Graduated Elastic Stockings on overall mortality at day 30 after randomization.

The secondary objective:

* To compare, in patients hospitalized for an acute medical illness, enoxaparin with Graduated Elastic Stockings versus enoxaparin placebo with Graduated Elastic Stockings on overall mortality at day 90 after randomization.
* To evaluate the safety of enoxaparin VTE prophylaxis in patients hospitalized for acute medical illness with respect to major hemorrhage, total bleedings, heparin induced thrombocytopenia, adverse events and serious adverse events .

ELIGIBILITY:
List of inclusion and exclusion criteria

Inclusion Criteria:

* Hospitalization within 48 hours prior randomization for at least one of the following medical acute medical illness:

  * Acute decompensation of heart failure
  * Severe systemic infection and at least one of the following:

    * Chronic pulmonary diseases (COPD, pulmonary fibrosis, pulmonary restrictive syndrome…)
    * Obesity (BMI ≥ 30kg/m2)
    * Personal history of VTE
    * Age ≥ 60 years
  * Active cancer (defined as being histologically confirmed with an initial diagnosis or recurrence or metastasis within the past 6 months) excluding planned hospitalization for chemotherapy
* Anticipated duration of hospitalization at least 6 days
* Health status:

  * ASA Health status score ≤ 3 (American Society of Anesthesiologists)
  * ECOG ≤ 2 in cancer patient
* Anticipated life expectancy > 1 week

Exclusion criteria:

* Major surgery or major trauma within the previous 6 weeks (orthopedic or trauma surgery to the lower extremities, gastrointestinal tract, urological, chest, gynecological surgery)
* Need for any ventilatory support (with intubation required)
* Symptomatic VTE at enrollment
* Multi organ failure
* Evidence of an active bleeding disorder
* Contraindication to anticoagulation:

  * Coagulopathy (acquired or inherited)
  * Neurosurgery within the past day 30
  * History of cerebral hemorrhage at any time
  * Known bacterial endocarditis
  * Uncontrolled arterial hypertension (systolic BP > 200 mmHg or diastolic BP > 110 mm Hg) at 2 successive readings
  * Haemostatic abnormalities: baseline platelet count <50,000/mm3, activated partial thromboplastin time (aPTT) 1.5x the upper limit of normal, or International Normalized Ratio (INR) > 1.5
  * Indication for thrombolytic therapy
  * Need for a curative treatment of anticoagulant therapy (low molecular weight heparin, unfractionated heparin, oral anticoagulant therapy)
  * Receiving LMWH or UFH at prophylactic doses for more than 72 hours prior to inclusion (patients receiving LMWH or UFH at prophylactic doses for 72 hours or less prior to entry may be included in the study)
  * Oral anticoagulant therapy within 72 hours prior to inclusion
* Cerebrovascular accident at inclusion and within 10 days prior study inclusion
* Prosthetic heart valves
* Confirmed cerebral metastases
* Known hypersensitivity to heparin or LMWH, or pork-derived products
* History of documented episode of heparin, or LMWH induced thrombocytopenia, and/or thrombosis (HIT, HAT, or HITTS)
* Participating in another clinical trial within the previous 30 days (patients with cancer included in a cancer treatment protocol are authorized to participate)
* Persistent renal failure (defined as a documented value of calculated creatinine clearance < 30 mL/min on at least 2 occasions ³3 days prior to entry into the study)
* Known or suspected severe anemia of unexplained cause considered clinically relevant by investigator
* Spinal or epidural analgesia or lumbar puncture within the preceding 24 hours
* Unlikely to be compliant (e.g. alcohol, drug abuse)
* Women of childbearing potential not protected by effective contraceptive method of birth control and/or who are unwilling to be tested for pregnancy (pregnancy status should be checked by serum or urine pregnancy testing prior to exposure to the investigational product)
* Refusal or inability to give informed consent to participate in the study
* Inability to be followed-up after discharge until day 90 after randomization

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8329 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Death rate with all causes mortality | At day 30
Hemorrhages | Occuring until day 90

SECONDARY OUTCOMES:
All-cause mortality | Between randomization and day 90
Adverse events, serious adverse events | During the entire observation period (from informed consent signature until Day 90)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno DESLANDES, Study Director — Sanofi
Locations (9):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Shanghai, China
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia

REFERENCES:
- [Derived] Kakkar AK, Cimminiello C, Goldhaber SZ, Parakh R, Wang C, Bergmann JF; LIFENOX Investigators. Low-molecular-weight heparin and mortality in acutely ill medical patients. N Engl J Med. 2011 Dec 29;365(26):2463-72. doi: 10.1056/NEJMoa1111288. PMID 22204723